CLINICAL TRIAL: NCT03015740
Title: Phase I/II Trial of MGCD516 Combined With Nivolumab in Patients With Advanced Clear Cell Renal Cell Cancer That Progressed on Prior VEGF-Targeted Therapy
Brief Title: Sitravatinib and Nivolumab in Treating Patients With Advanced or Metastatic Kidney Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0332; NCI-2017-00324 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0332 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Clear Cell Renal Cell Carcinoma; Metastatic Kidney Carcinoma; Stage III Renal Cell Cancer AJCC v7; Stage IV Renal Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab; sitravatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (sitravatinib, nivolumab) (Experimental): Patients receive sitravatinib PO QD on days 1-14 and receive nivolumab IV over 60 minutes on day 1 starting cycle 2. Cycles repeat every 14 days for cycles 1-6 and then every 28 days for subsequent cycles in the absence of disease progression or unacceptable toxicity. Patients who receive at least 6 infusions of nivolumab with no DLTs related to nivolumab, may then receive nivolumab every 4 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Sitravatinib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Sitravatinib — Given PO
  Other Names: MGCD516

SUMMARY:
This phase I/II trial studies the side effects of sitravatinib and how well it works with nivolumab in treating patients with kidney cancer that has spread to other places in the body. Sitravatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving sitravatinib and nivolumab may work better in treating patients with kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the toxicities (defined as a grade 3 or 4 National Cancer Institute [NCI] non-hematologic or hematologic adverse event, within 12 weeks from treatment initiation), and efficacy (defined as achieving complete remission, partial remission, or stable disease within 6 weeks) of sitravatinib (MGCD516) when administered orally (PO) daily in combination with standard dose nivolumab 240 mg/kg every 2 weeks.

SECONDARY OBJECTIVES:

I. To estimate the overall survival (OS), progression-free survival (PFS) times, objective response rates (ORR), and quality of life (QOL) of patients with advanced clear cell renal cell cancer (RCC) treated with the combination of MGCD516 and nivolumab.

II. Evaluate potential biomarkers for patient stratification and treatment response, including genetic analysis, serum cytokines and chemokines, as well as tumor antigen-specific immune responses, such as antibody and T cell responses, as surrogates for anti-tumor activity.

OUTLINE:

Patients receive sitravatinib PO once daily (QD) on days 1-14 and receive nivolumab intravenously (IV) over 60 minutes on day 1 starting cycle 2. Cycles repeat every 14 days for cycles 1-6 and then every 28 days for subsequent cycles in the absence of disease progression or unacceptable toxicity. Patients who receive at least 6 infusions of nivolumab with no dose limiting toxicities (DLTs) related to nivolumab, may then receive nivolumab every 4 weeks.

After completion of study treatment, patients are followed up at 30 days and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed metastatic/advanced clear cell RCC, or RCC with a clear cell component, who have received 1 or 2 prior anti-angiogenic therapy regimens (+/- cytokine therapy with interleukin-2 or interferon-alfa) in the advanced or metastatic setting; examples of anti-angiogenic agents include, but are not limited to, sorafenib, sunitinib, pazopanib, axitinib, and bevacizumab
* There must be evidence of progression on or after last treatment regimen received and within 6 months of enrollment
* Patients must have at least one measurable site of disease, defined as a lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) and measures >= 15 mm with conventional techniques or >= 10 mm with more sensitive techniques such as magnetic resonance imaging (MRI) or spiral computed tomography (CT) scan; if the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation
* Karnofsky performance status >= 70
* Hemoglobin >= 9 g/dl (treatment allowed) (within 14 days prior to study entry)
* Absolute neutrophil count >= 1,500/uL (within 14 days prior to study entry)
* Platelets >= 100,000/uL (within 14 days prior to study entry)
* Total bilirubin =< 1.5 mg/dl (within 14 days prior to study entry)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) or alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (ULN), except in known hepatic metastasis, wherein may be < 5 x ULN (within 14 days prior to study entry)
* Serum creatinine =< 1.5 x ULN (as long as patient does not require dialysis); a) may receive transfusion b) if creatinine is not < 1.5 x ULN, then calculate by Cockcroft-Gault methods or local institutional standard and creatinine clearance (CrCl) must be >= 40 mL/kg/1.73 m^2 (within 14 days prior to study entry)
* International normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 x ULN within 14 days prior to study entry; therapeutic anticoagulation with warfarin is allowed if target INR =< 3 on a stable dose of warfarin or on a stable dose of low molecular weight (LMW) heparin for > 2 weeks (14 days) at the time of enrollment
* Female patients of childbearing potential (not postmenopausal for at least 12 months and not surgically sterile) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 14 days before study entry; pregnancy test must be repeated if performed > 14 days before starting study drug
* Women must not be breastfeeding
* Patients with a history of major psychiatric illness must be judged (by the treating physician) able to fully understand the investigational nature of the study and the risks associated with the therapy
* Patients with controlled brain metastases are allowed on protocol if they had solitary brain metastases that was surgically resected or treated with radiosurgery or gamma knife, without recurrence or edema for 1 month (4 weeks)

Exclusion Criteria:

* Patients must not have any other malignancies within the past 2 years except for in situ carcinoma of any site, or adequately treated (without recurrence post-resection or post-radiotherapy) carcinoma of the cervix or basal or squamous cell carcinomas of the skin or active non-threatening second malignancy that would not, in the investigator's opinion, potentially interfere with the patient's ability to participate and/or complete this trial; examples include but not limited to: urothelial cancer grade Ta or T1, adenocarcinoma of the prostate treated by active surveillance
* Patients currently receiving anticancer therapies or who have received anticancer therapies within 2 weeks (14 days) from enrollment into this study (including chemotherapy and targeted therapy) are excluded; also, patients who have completed palliative radiation therapy more than 14 days prior to the first dose of MGCD516 are eligible
* Patients, who have had a major surgery or significant traumatic injury (injury requiring > 4 weeks [28 days] to heal) within 4 weeks (28 days) of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that are expected to require major surgery during the course of the study
* Patients who have been previously treated with mTOR inhibitors such as everolimus and temsirolimus, or with c-MET inhibitors such as cabozantinib
* Patients who have organ allografts
* Known or suspected autoimmune disease; patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) and autoimmune disorders such as rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus or autoimmune vasculitis (e.g., Wegener's granulomatosis) are excluded from this study; patients with a history of Hashimoto's thyroiditis only requiring hormone replacement, type I diabetes, or psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are allowed to participate
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Any underlying medical condition, which in the opinion of the investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events, such as a condition associated with frequent diarrhea, uncontrolled nausea, vomiting, malabsorption syndrome or small bowel resection that may significantly alter the absorption of MGCD516
* Patients must not have received prior anticancer therapy with any immune checkpoint inhibitors such as anti-CLTA-4, anti-PD1, or anti-PD-L1
* Patients receiving any concomitant systemic therapy for renal cell cancer are excluded
* Patients must not be scheduled to receive another experimental drug while on this study
* Patients who are on high dose steroid (e.g., > 10 mg prednisone daily or equivalent) or other more potent immune suppression medications (e.g., infliximab); topical, inhaled, intra-articular, ocular, or intranasal corticosteroids (with minimal systemic absorption) are allowed; a brief course (=< 48 hours) of systemic corticosteroids for prophylaxis (e.g., from contrast dye allergy) is permitted
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as: symptomatic congestive heart failure of New York Heart Association class III or IV; unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease; severely impaired lung function as defined as oxygen (O2) saturation that is 88% or less at rest on room air; uncontrolled diabetes as defined by blood glucose > 200 mg/dl (11.1 mmol/l); systemic fungal, bacterial, viral, or other infection that is not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement) despite appropriate antibiotics or other treatment; liver disease such as cirrhosis or chronic active hepatitis; positive test for hepatitis B virus (HBV) using HBV surface antigen (HBV sAg) test or positive test for hepatitis C virus (HCV) using HCV ribonucleic acid (RNA) or HCV antibody test indicating acute or chronic infection
* Patients must not have history of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of MGCD516 or nivolumab or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications
* Patients should not receive immunization with attenuated live vaccines within one week (7 days) of study entry or during study period
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods; if barrier contraceptives are being used, these must be continued throughout the trial by both sexes; hormonal contraceptives are not acceptable as a sole method of contraception; (women of childbearing potential must have a negative urine or serum pregnancy test within 14 days prior to study entry; pregnancy test must be repeated if performed > 14 days before administration of MGCD516)
* Any patients who cannot be compliant with the appointments required in this protocol must not be enrolled in this study
* Concurrent therapy with medications known to significantly prolong the QT interval and/or associated with increased risk for Torsade de Pointes arrhythmia; the principal investigator (PI) is the final arbiter in questions related to eligibility
* Patients with left ventricular ejection fraction (LVEF) < 40%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-04-23 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavlos Msaoel, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April 2017 to February 2020, patients were recruited from the outpatient clinics for Genitourinary Medical Oncology at MD Anderson Cancer Center in Houston, Texas who have been diagnosed with cancer and currently undergoing outpatient treatment at the cancer center that are immunotherapy-naïve with ccRCC refractory to prior antiangiogenic therapies.
Pre-assignment Details: 42 participants were randomized on trial
Groups:
- Received Sitravatinib 80 mg in Combination With Nivolumab: combination of sitravatinib 80 MG and the anti-PD-1 agent nivolumab
- Received Sitravatinib 120 mg in Combination With Nivolumab: combination of sitravatinib 120 MG and the anti-PD-1 agent nivolumab
- Received Sitravatinib 150 mg in Combination With Nivolumab: combination of sitravatinib 150 MG and the anti-PD-1 agent nivolumab
Period: Overall Study
Arm/Group | Received Sitravatinib 80 mg in Combination With Nivolumab | Received Sitravatinib 120 mg in Combination With Nivolumab | Received Sitravatinib 150 mg in Combination With Nivolumab
Started | 15 | 24 | 3
Completed | 9 | 19 | 3
Not Completed | 6 | 5 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Death | 3 | 5 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Dosed participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Received Sitravatinib 80 mg in Combination With Nivolumab | Received Sitravatinib 120 mg in Combination With Nivolumab | Received Sitravatinib 150 mg in Combination With Nivolumab | Total
Number analyzed (Participants) | 15 | 24 | 3 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 10 | 3 | 17
  >=65 years | 11 | 14 | 0 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 0 | 7
  Male | 13 | 19 | 3 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 0 | 4
  Not Hispanic or Latino | 11 | 23 | 3 | 37
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 12 | 21 | 3 | 36
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 24 | 3 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: To determine the toxicities (defined as a grade 3 or 4 National Cancer Institute [NCI] non-hematologic or hematologic adverse event, within 12 weeks from treatment initiation),and efficacy (defined as achieving complete remission, partial remission, or stable disease within 6 weeks) of dosing.
Time Frame: from enrollment up to 12 weeks for each dosing group
Population: A participant is considered enrolled when study medication is administered on Day 1
Measure: Number; unit: participants
Groups:
- Received Sitravatinib 80 mg in Combination With Nivolumab: combination of sitravatinib and the anti-PD-1 agent nivolumab
Arm/Group | Received Sitravatinib 80 mg in Combination With Nivolumab | Received Sitravatinib 120 mg in Combination With Nivolumab | Received Sitravatinib 150 mg in Combination With Nivolumab
Number analyzed (Participants) | 15 | 24 | 3
participants
  DLTs within 12 weeks | 4 | 10 | 3
  disease control at 6 weeks | 13 | 21 | 3

2. Secondary Outcome: Overall Survival (OS)
Description: To estimate the overall survival (OS) of patients with advanced clear cell renal cell cancer (RCC) treated with the combination of MGCD516 and nivolumab. The Secondary objective of the protocol is to capture combined results from all subjects who received treatment of the combination therapy. The intent was not to report results for each arm/group.
Time Frame: From enrollment to study completion, up to 5 years 4 months
Measure: Count of Participants; unit: Participants
Groups:
- Received Sitravatinib (MGCD516) Combined With Nivolumab: combination of sitravatinib and the anti-PD-1 agent nivolumab
Arm/Group | Received Sitravatinib (MGCD516) Combined With Nivolumab
Number analyzed (Participants) | 42
Participants | 34

3. Secondary Outcome: Progression-free Survival (PFS) Times
Description: To estimate the progression-free survival (PFS) times of patients with advanced clear cell renal cell cancer (RCC) treated with the combination of MGCD516 and nivolumab. : The Secondary objective of the protocol is to capture combined results from all subjects who received treatment of the combination therapy. The intent was not to report results for each arm/group.
Time Frame: From enrollment to study completion, up to 5 years 4 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Received Sitravatinib (MGCD516) Combined With Nivolumab
Number analyzed (Participants) | 42
months | 11.7 [8.2 to 16.6]

4. Secondary Outcome: Objective Response Rates (ORR)
Description: To estimate the objective response rates (ORR) of patients with advanced clear cell renal cell cancer (RCC) treated with the combination of MGCD516 and nivolumab. The Secondary objective of the protocol is to capture combined results from all subjects who received treatment of the combination therapy. The intent was not to report results for each arm/group.
Time Frame: From enrollment to study completion, up to 5 years 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Received Sitravatinib (MGCD516) Combined With Nivolumab
Number analyzed (Participants) | 42
Participants | 15

ADVERSE EVENTS:
Time Frame: up to 5 years and 4 months
Description: Death A life-threatening adverse drug experience - any adverse experience that places the patient, in the view of the initial reporter, at immediate risk of death from the adverse experience as it occurred. It does not include experience that, had it occurred in a more severe form, might have caused death.
Arm/Group | Received Sitravatinib 80 mg in Combination With Nivolumab | Received Sitravatinib 120 mg in Combination With Nivolumab | Received Sitravatinib 150 mg in Combination With Nivolumab
All-Cause Mortality (participants affected / at risk) | 3/15 | 5/24 | 0/3
Serious Adverse Events (participants affected / at risk) | 8/15 | 14/24 | 2/3
Other Adverse Events (participants affected / at risk) | 13/15 | 23/24 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Received Sitravatinib 80 mg in Combination With Nivolumab (N=15) | Received Sitravatinib 120 mg in Combination With Nivolumab (N=24) | Received Sitravatinib 150 mg in Combination With Nivolumab (N=3)
abodominal pain (Gastrointestinal disorders) | 1 | 0 | 0
acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
appendicitus (Infections and infestations) | 1 | 1 | 0
bronchial obsturction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
creatinine increased (Investigations) | 0 | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0 | 0 — GI Bleed
Hematoma (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Myasthenia Gravis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Portal vein thrombosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Sudden death NOS (General disorders) | 0 | 1 | 0
Surgical and medical procedures - Other, specify (Gastrointestinal disorders) | 0 | 1 | 0 — Disc Removal Surgery
Surgical and medical procedures - Other, specify (General disorders) | 1 | 0 | 1 — Cryoplasty and Vertebroplasty to T1 and T3
Surgical and medical procedures - Other, specify (General disorders) | 1 | 0 | 1 — Pain Control After IR Procedure
Surgical and medical procedures - Other, specify (nephrectomy in conjunction with hepatectomy) (Renal and urinary disorders) | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 2 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vertigo (General disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Received Sitravatinib 80 mg in Combination With Nivolumab (N=15) | Received Sitravatinib 120 mg in Combination With Nivolumab (N=24) | Received Sitravatinib 150 mg in Combination With Nivolumab (N=3)
Anemia (Blood and lymphatic system disorders) | 13 | 21 | 2
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 3 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 2 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 4 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 3 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 0 | 2
Ear pain (Ear and labyrinth disorders) | 2 | 1 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0
Endocrine disorders - Other, specify (Endocrine disorders) | 5 | 6 | 3
Hyperthyroidism (Endocrine disorders) | 1 | 2 | 1
Hypothyroidism (Endocrine disorders) | 4 | 14 | 3
Blurred vision (Eye disorders) | 1 | 6 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 0
Eye disorders - Other, specify (Eye disorders) | 0 | 2 | 0
Flashing lights (Eye disorders) | 0 | 0 | 1
Watering eyes (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 9 | 2
Bloating (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 8 | 14 | 1
Diarrhea (Gastrointestinal disorders) | 11 | 22 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 | 3 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 6 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 12 | 2
Oral dysesthesia (Gastrointestinal disorders) | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 1 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 7 | 5 | 2
Chills (General disorders) | 2 | 0 | 0
Edema Limbs (General disorders) | 5 | 9 | 0
Edema trunk (General disorders) | 0 | 1 | 0
Facial pain (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 12 | 23 | 3
Fever (General disorders) | 3 | 3 | 0
Flu like symptoms (General disorders) | 2 | 0 | 1
Gait disturbance (General disorders) | 2 | 4 | 0
Irritability (General disorders) | 1 | 0 | 0
Localized edema (General disorders) | 1 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 4 | 0
Pain (General disorders) | 6 | 8 | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 | 5 | 2
Anorectal infection (Infections and infestations) | 0 | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 1 | 0
Sinusitis (Infections and infestations) | 4 | 2 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 0
Bruising (Injury, poisoning and procedural complications) | 3 | 2 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 3 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 5 | 2 | 1
Alanine aminotransferase increased (Investigations) | 7 | 21 | 3
Alkaline phosphatase increased (Investigations) | 5 | 13 | 1
Aspartate aminotransferase increased (Investigations) | 6 | 19 | 2
Blood bilirubin increased (Investigations) | 2 | 3 | 0
Cardiac troponin I increased (Investigations) | 1 | 0 | 0
Cholesterol high (Investigations) | 7 | 20 | 3
Creatinine increased (Investigations) | 12 | 20 | 3
Hemoglobin increased (Investigations) | 1 | 1 | 0
INR increased (Investigations) | 5 | 2 | 0
Investigations - Other, specify (Investigations) | 12 | 23 | 3
Lipase increased (Investigations) | 11 | 15 | 1
Lymphocyte count decreased (Investigations) | 10 | 7 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 2 | 9 | 0
Serum amylase increased (Investigations) | 10 | 12 | 2
Weight gain (Investigations) | 0 | 1 | 1
Weight loss (Investigations) | 12 | 13 | 2
White blood cell decreased (Investigations) | 2 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 11 | 17 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 4 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 13 | 23 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 7 | 9 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypernatremia (Metabolism and nutrition disorders) | 2 | 4 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 13 | 17 | 3
Hypoalbuminemia (Investigations) | 6 | 9 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 3 | 0
Hypoglycemia (Investigations) | 2 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 6 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 5 | 0
Hyponatremia (Metabolism and nutrition disorders) | 5 | 11 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 15 | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 5 | 7 | 2
Concentration impairment (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 5 | 8 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 1
Dysphasia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 5 | 11 | 3
Hypersomnia (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 2 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 2 | 0
Paresthesia (Nervous system disorders) | 2 | 5 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3 | 0
Sinus pain (Nervous system disorders) | 0 | 4 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Vasovagal reaction (Nervous system disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 9 | 2
Confusion (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 2 | 1
Insomnia (Psychiatric disorders) | 5 | 8 | 2
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 4 | 0
Hematuria (Renal and urinary disorders) | 1 | 9 | 0
Proteinuria (Renal and urinary disorders) | 10 | 20 | 2
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 | 8 | 1
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Urinary frequency (Renal and urinary disorders) | 3 | 3 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 10 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 18 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 13 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 7 | 11 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 11 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 5 | 10 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 2
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 5 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 9 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 9 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 7 | 5 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 7 | 3
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 | 6 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 2 | 3 | 1
Hot flashes (Vascular disorders) | 1 | 4 | 1
Hypertension (Vascular disorders) | 9 | 20 | 2
Lymphocele (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 2 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 13 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 15 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 6 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 9 | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT03015740/Prot_SAP_000.pdf